CLINICAL TRIAL: NCT02978352
Title: A Comparison of Learning Effectiveness of Confusion Assessment Method (CAM-ICU) Between E-learning and Conventional Face-to-face Lecture and Demonstration
Brief Title: A Comparison of Learning Method (CAM-ICU) Between E-learning and Conventional Face-to-face Lecture and Demonstration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 300/2559(EC4)
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- face-to-face (Experimental): Traditional learning group (face-to-face): 4 different sessions will be conducted to suit the participants' convenience Duration of each session is 60-90 minutes Each session comprises lecture, video demonstration of CAM-ICU assessment, discussion, volunteer participation during class demonstration
  Interventions: Other: learning
- E-learning (Experimental): 60-90 minute online course will be accessible through intranet Wi-Fi The course encompasses types, incidence, risk factors, significance and effects of delirium, diagnostic criteria and CAM-ICU application Inclusion of video demonstration of simulated patients and CAM-ICU application, common pitfalls of healthcare providers, and practice questions
  Interventions: Other: learning

INTERVENTIONS:
Other: learning

SUMMARY:
Delirium is an acute and fluctuating disturbance of consciousness characterized by reduced attention, impaired cognition and perception, usually resulting from general physical conditions. Delirium contributes to longer hospital length of stay, increased mortality, increased healthcare costs, and long-term cognitive and functional impairment. However, it is often underdiagnosed and undertreated. E-learning (electronic learning) proves to be a time-efficient, flexible and convenient training method, making it suitable for a large organization like Siriraj hospital where there is a large employee turnover rate. So the investigators want to compare the passing rate between the e-learning group and the traditional learning group.

DETAILED DESCRIPTION:
Primary objective: Compare the passing rate between the e-learning group and the traditional learning group

Secondary objectives: Assess the trainees' satisfaction and problems associated with e-learning implementation, Investigate the causes of inaccurate CAM-ICU assessment for improvement in future training sessions

ELIGIBILITY:
Inclusion Criteria:

* ICU nurse
* general ward nurse
* private ward nurses
* nurse anesthetists

Exclusion Criteria:

* Previous exposure to CAM-ICU
* Inability to complete the training courses
* Inability to complete the required 3 simulated patient scenarios

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The passing rate between the e-learning group and the traditional learning group | 2 weeks

SECONDARY OUTCOMES:
Assess the trainees' satisfaction | 2 weeks
  Satisfaction score from 0 (dissatisfy) and 10 (very satisfy)
Investigate the causes of inaccurate CAM-ICU assessment for improvement in future training sessions | 2 weeks

IPD SHARING:
Plan to Share IPD: No